CLINICAL TRIAL: NCT05803343
Title: Evaluating Additive Effects of Including Canines in Regulating Together: A Group Treatment to Address Emotion Dysregulation in Youth With Autism Spectrum Disorder
Brief Title: Evaluating Additive Effects of Including Canines in Regulating Together
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01HD106353 (NIH)
Record Dates: First submitted 2023-03-15; First posted 2023-04-07 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Autism Spectrum Disorder; Emotion Regulation
MeSH Terms: conditions — Autism Spectrum Disorder; Emotional Regulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regulating Together-Canine (RT-Canine) (Experimental): Participants in this Arm will receive the Regulating Together-Canine intervention.
  Interventions: Behavioral: Regulating Together-Canine
- Regulating Together-Standard (RT-Standard) (Active Comparator): Participants in this Arm will receive the Regulating Together-Standard intervention.
  Interventions: Behavioral: Regulating Together-Standard

INTERVENTIONS:
Behavioral: Regulating Together-Canine — RT-C is an animal assisted, intensive outpatient group intervention for children with autism spectrum disorder and emotion dysregulation. RT-C meets for 1.5 hours, twice weekly for five weeks with concurrent youth and caregiver groups. The children progress through skills including relaxation training, arousal ratings, problem size, mindfulness, problem solving, and cognitive flexibility. The caregivers learn crisis management, reward systems, and coaching strategies for topics taught to the children. Homework is utilized to reinforce use of skills outside the group. The canines are present throughout as both a calming presence and teaching assistant. Children will be able to interact with the dog when practicing relaxation at the beginning of each session and throughout the session. Additionally, the dog will help to emphasize certain curriculum concepts.
  Other Names: RT-Canine, RT-C
  Arms: Regulating Together-Canine (RT-Canine)
Behavioral: Regulating Together-Standard — RT-S an established, intensive outpatient group intervention for children with autism spectrum disorder and emotion dysregulation. It engages both caregivers and children and utilizes evidence-based intervention techniques including cognitive behavioral therapy (CBT), visuals, reinforcements, and scaffolding, and newer interventions such as mindfulness and acceptance-based therapy.
  Other Names: RT-Standard, RT-S
  Arms: Regulating Together-Standard (RT-Standard)

SUMMARY:
The primary objective is to evaluate the potential additive effect of animal-assisted intervention (AAI) on a manualized behavioral treatment targeting emotion dysregulation (ED) in children with autism spectrum disorder (ASD).

Aim 1: Evaluate whether Regulating Together-Canine demonstrates earlier and greater improvement in emotion dysregulation than Regulating Together-Standard.

Aim 2: Evaluate if Regulating Together-Canine increases child engagement and learning compared to Regulating Together-Standard.

Exploratory Aim: Explore association of physiological arousal (via heart rate tracking) with emotion dysregulation, treatment engagement, and learning.

DETAILED DESCRIPTION:
Children between the ages of 8 years 0 months and 15 years 11 months with Autism Spectrum Disorder (ASD) and emotion dysregulation (ED) and their caregivers will participate in 5 research visits and 10 group intervention sessions. They are randomly assigned to either Regulating Together-Standard group (no dog), or Regulating Together-Canine group (with dog). Characterization measures will be completed at Screen (T1). All outcome measures will be completed at Baseline (T2), Post-treatment (1-2 weeks following treatment completion, T3), 10 week post treatment completion follow up (T4), and 6 month post treatment completion follow up (T5).

ELIGIBILITY:
Inclusion Criteria:

* Concern of emotion dysregulation (ED) as measured by a score of 6 or greater on the Emotion Dysregulation Inventory-Reactivity (EDI-R)
* Diagnosis of autism spectrum disorder (ASD)
* Diagnosis confirmed by an experienced ASD clinician and further supported by scoring in the range for ASD on the Autism Diagnostic Observation Schedule (ADOS-2)
* A Full Scale Intelligence Quotient score of 65 or greater on the Weschler Abbreviated Scale Intelligence (WASI-II)
* English is the primary language
* Family willing to keep prescribed medication stable over the course of the study period

Exclusion Criteria:

* Participant has a phobia toward or is allergic to canines
* Participant has a history of aggression toward animals
* Participant has had any physical aggression toward other children outside the home in the past 2 weeks that resulted in injury
* Presence of comorbid major neuropsychiatric illness warranting other treatment approaches as determined by the study clinician(s) including substance use disorders, psychotic disorders/schizophrenia, and bipolar disorder, among others
* Presence of any major sensory impairment that would limit participating in the material including blindness or uncorrected hearing loss
* A legal guardian is not available to provide informed consent

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Emotion Dysregulation Inventory-Reactivity (EDI-R) | Through study completion
  The EDI-R is a parent-report measure that consists of two scales, Reactivity which captures poorly regulated negative emotional responses and Dysphoria characterized by decreased uptake of positive affect and lack of motivation. Higher scores indicate higher emotional reactivity.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Shaffer, Psy.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States